CLINICAL TRIAL: NCT06430424
Title: Study of Metabolic, Genomic and Proteomic Modifications in Relapsed Glioblastoma. Identification or Prognostic Markers in Patients Undergoing Surgery for Relapsed Glioblastoma.
Brief Title: Study of Metabolic, Transcriptomic and Proteomic Characteristics in Relapsed Glioblastoma
Acronym: GBrecurr
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/79
Record Dates: First submitted 2024-03-27; First posted 2024-05-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Relapsed Cancer; Glioblastoma IDH (Isocitrate Dehydrogenase) Wildtype
Keywords: Recurrent glioblastoma; Prognostic; Metabolism; Proteomic; Transcriptomic; Microbiota
MeSH Terms: conditions — Recurrence; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients operated for primary and recurrent glioblastoma: Patients operated for both primary and recurrent glioblastoma between 2005 and 2023 at the CHU de Bordeaux
  Interventions: Biological: Relapsed glioblastoma

INTERVENTIONS:
Biological: Relapsed glioblastoma — Paired tumor samples diagnosis/relapse

SUMMARY:
Glioblastomas are the most frequent and aggressive malignant tumors of the CNS in adults, with almost systematic relapse despite treatment with surgery followed by radio-chemotherapy (STUPP protocol). The aim of this study is to better characterize transcriptomic, proteomic and metabolic changes in relapsed glioblastoma compared to the initial tumor, in order to identify new prognostic markers and potential new therapeutic targets.

DETAILED DESCRIPTION:
Glioblastomas are the most frequent and aggressive malignant Central Nervous System (CNS) tumors in adults, with a median survival of only 14 months.

Current treatment is based on surgery followed by radiochemotherapy (STUPP protocol), unchanged since 2005. Clinical trials evaluating immune checkpoint inhibitors and targeted therapies have largely failed to demonstrate efficacy in these tumors. In order to better understand the oncogenesis of glioblastoma and identify potential new therapeutic targets, the study of the characteristics of relapsed tumors compared with the initial tumor seems relevant.

The aim of this retrospective study is to investigate the transcriptomic, proteomic and metabolic characteristics of relapsed glioblastomas reoperated at the University Hospital of Bordeaux, France, between 2005 and 2023, for which tumor material is available. These analyses will be correlated with relapse-free and overall survival of the patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* surgery for both primary and recurrent glioblastoma between 2005 and 2023 at the CHU de Bordeaux

Exclusion Criteria:

* systemic therapy received for non-glioblastoma tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed glioblastomas reoperated at the University Hospital of Bordeaux, France, between 2005 and 2023, for which tumor material is available
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of metabolic changes involved in glioblastoma relapse | Up to 2 years after the start of the study
  Relative abondance of metabolite and differential enzyme expression in a recurrence versus primary sample

SECONDARY OUTCOMES:
Progression-free survival | From date of the second surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  Progression-free survival of patients who underwent surgery for relapse glioblastoma after the surgery of relapse measured at time of inclusion
Overall survival | From date of the second surgery until the date of death from any cause, assessed up to 5 years
  Overall survival of patients who underwent surgery for relapse glioblastoma after the surgery of relapse

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux - Hôpital Saint-André, Service d'Oncologie Médicale, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No